CLINICAL TRIAL: NCT06890754
Title: Performance of Hysteroscopy in Diagnosing Chronic Endometritis and the Role of Intra- and Inter-Observer Variability: A Prospective Study of 70 Cases.
Brief Title: Hysteroscopy for Chronic Endometritis: Diagnostic Performance and Observer Variability
Status: Completed | Type: Observational
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Haithem Aloui, university hospital assistant, Tunis University
Other Study IDs: Endometrite hysteroscopy
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Endometritis
Keywords: Chronic endometritis; intra-observer variability; inter-observer variability; hysteroscopy; CD138
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic hysteroscopy — Diagnostic hysteroscopy. An IHC study of the expression of the plasma cell marker CD138 was systematically performed for all samples studied

SUMMARY:
This study investigates the role of hysteroscopy in diagnosing chronic endometritis (CE), a condition linked to female infertility but difficult to diagnose due to nonspecific symptoms. While histological examination with CD138 ( Cluster of Differentiation 138 )immunohistochemistry is the gold standard, hysteroscopy remains widely used. This prospective, multicenter study included infertile women with no uterine abnormalities on ultrasound. Hysteroscopy was performed using standardized criteria, and its diagnostic performance was compared to histopathology. Intra- and inter-observer variability were also assessed through blinded video evaluations by two specialists. The study aimed to determine the reliability of hysteroscopy in diagnosing CE and its agreement among different observers.

DETAILED DESCRIPTION:
This study evaluates the diagnostic performance of hysteroscopy in detecting chronic endometritis (CE), a condition associated with female infertility. CE is characterized by persistent endometrial inflammation and is challenging to diagnose due to its nonspecific clinical presentation. Histopathological examination with CD138 immunohistochemistry (IHC) is currently the gold standard for CE diagnosis, yet hysteroscopy remains a commonly used tool in clinical practice.

This prospective, multicenter study was conducted between June 6, 2021, and August 8, 2022, and included infertile women aged 18 to 42 years. Participants were selected based on normal pelvic ultrasound findings, while patients with biological inflammatory syndrome, recent acute genital infections, autolysed biopsies, unusable hysteroscopy videos, atypical hyperplasia, or endometrial cancer were excluded. The final cohort comprised 70 patients.

Hysteroscopy was performed during the late follicular phase (days 8-12) using a 2.9 mm 30° rigid hysteroscope with saline distension. The procedure was conducted using a "no-touch" technique to minimize endometrial trauma and ensure accurate video interpretation. Endometrial biopsies were obtained using a Novak curette for subsequent CD138 IHC analysis.

The hysteroscopic diagnosis of CE was based on standardized criteria proposed by Cicinelli et al., including micro polyps, focal and diffuse hyperaemia, stromal oedema, strawberry aspect, and haemorrhagic spots. Recorded hysteroscopic videos were independently reviewed by two reproductive medicine specialists. To assess intra- and inter-observer variability, a second blinded evaluation was conducted four weeks later by the same observers.

The study aimed to assess the sensitivity, specificity, and predictive values of hysteroscopy in diagnosing CE while evaluating the consistency of observer interpretations. By comparing hysteroscopic findings to histopathological results, the study provides insights into the reliability of hysteroscopy as a diagnostic tool for CE and highlights its limitations due to observer variability.

ELIGIBILITY:
Inclusion Criteria:

* included women aged 18 to 42 years, consulting for infertility, with a pelvic ultrasound showing no uterine abnormalities

Exclusion Criteria:

* Excluded from the study were patients with biological inflammatory syndrome, those on antibiotic therapy or with a recent acute genital infection (less than three months), autolysed biopsies, unusable hysteroscopy videos, atypical hyperplasia, or endometrial cancer.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consisted of infertile women aged 18 to 42 years with no uterine abnormalities on pelvic ultrasound. Exclusion criteria included biological inflammatory syndrome, recent acute genital infections (within three months), antibiotic therapy, autolysed biopsies, unusable hysteroscopy videos, atypical hyperplasia, and endometrial cancer. The sample size was determined based on the reported prevalence of chronic endometritis (CE) in infertile women, ranging from 2.8% to 30%, with a calculated target of 68 participants to ensure statistical significance at a 95% confidence level.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Undergoing Diagnostic Hysteroscopy | peroperatively
  Examination of the uterine cavity and the cervico-isthmic canal.
Expression of CD138 Marker in Endometrial Biopsy | First 24 hours
  An immunohistochemical study of plasma cell marker CD138 expression was systematically performed on all analyzed samples. The anti-CD138 monoclonal antibody (Clone Ml15, Leica Biosystems, Reference: PA0088), ready to use on the BOND immunohistochemistry automated system, was used.

CONTACTS AND LOCATIONS:
Overall Officials: Haithem Aloui, Principal Investigator — Tunis University Manar
Locations (1):
- Haithem Aloui, Manouba, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No
This study's individual participant data (IPD) will be made available to researchers upon reasonable request. The shared data will include de-identified participant-level datasets containing:
  Demographic characteristics (age, Body Mass Index, smoking status, infertility duration, primary versus secondary infertility) Hysteroscopic findings (micro polyps, focal hyperaemia, diffuse hyperaemia, stromal oedema, strawberry aspect, haemorrhagic spots) Histopathological results (CD138, immunohistochemistry findings, plasma cell count per high-power field) Observer assessments (initial and repeat evaluations for intra- and inter-observer variability) All data will be de-identified to ensure confidentiality. Access will be granted to qualified researchers for meta-analyses, systematic reviews, or investigations related to chronic endometritis and infertility, following approval of a research proposal and data-sharing agreement.